CLINICAL TRIAL: NCT04558515
Title: Clinical Evaluation of Automated Microscope Solutions for Malaria Diagnosis
Brief Title: Automated Microscopy Evaluation Study
Acronym: AutoMic
Status: Completed | Type: Observational
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: MA013
Record Dates: First submitted 2020-09-15; First posted 2020-09-22 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Symptomatic patients positive for malaria by PCR
  Interventions: Diagnostic Test: Novel malaria diagnostics & tools
- Control: Symptomatic patients negative for malaria by PCR
  Interventions: Diagnostic Test: Novel malaria diagnostics & tools

INTERVENTIONS:
Diagnostic Test: Novel malaria diagnostics & tools — Next generation microscopy tools for malaria diagnosis and medical applications

SUMMARY:
Since the introduction of Giemsa stain in 1904 until today, malaria microscopy has been the standard of practice for malaria diagnosis. However, microscopic detection of malaria parasites is labour-intensive, time-consuming and expertise-demanding. Moreover, the slide interpretation is highly dependent on the staining technique and the technician's expertise.

To address these, multiple organisations have developed next generation microscopes to move towards a next generation microscope that can improve slide preparation, interpretation or data collection, or a combination of these features.

In this study, a prospective evaluation of miLab™ and other next generation automated microscope solutions as well as a malaria rapid diagnostic test (RDT) reader app will be performed in malaria-endemic countries to assess their clinical performance for detection of malaria clinical cases at POC.

ELIGIBILITY:
Inclusion Criteria:

* Aged 5 years or older
* Malaria status (positive or negative) established by microscopy at the health facility, where the patient is presenting
* Freely agreeing to participate by signing an informed consent form (adults aged 18 and older and parent/legal guardian of a child) and providing assent (children aged 13-17)
* Willing to provide finger prick blood sample at enrollment

Exclusion Criteria:

* Having received antimalarial treatment during the preceding four-week period
* Presence of symptoms and signs of severe disease and/or central nervous system infections, as defined by WHO guidelines

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with symptoms suggestive of malaria seeking clinical care in health facilities
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical performance assessment | up to 6 months
  Point estimates of clinical performance characteristics with 95% confidence intervals (sensitivity, specificity) of next generation microscopy tools using nPCR as the reference test for the detection of malaria clinical cases
Concordance | up to 6 months
  Point estimate with 95% confidence intervals of the percentage agreement in interpreting malaria diagnostics between the app and visual reading

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Endemic Diseases, Medical Campus, Khartoum, Sudan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hamid MMA, Mohamed AO, Mohammed FO, Elaagip A, Mustafa SA, Elfaki T, Jebreel WMA, Albsheer MM, Dittrich S, Owusu EDA, Yerlikaya S. Diagnostic accuracy of an automated microscope solution (miLab) in detecting malaria parasites in symptomatic patients at point-of-care in Sudan: a case-control study. Malar J. 2024 Jun 28;23(1):200. doi: 10.1186/s12936-024-05029-3. PMID 38943203